CLINICAL TRIAL: NCT01991587
Title: Safety, Tolerability and Immunogenicity of a Plant-made Seasonal Quadrivalent Virus-like-particle (VLP) Influenza Vaccine in Adults
Brief Title: Safety, Tolerability and Immunogenicity of a Plant-made Seasonal Quadrivalent VLP Influenza Vaccine in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-Q12VLP-004
Record Dates: First submitted 2013-11-06; First posted 2013-11-25 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2019-11

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Influenza; Human; RNA Virus Infections; Immunologic; Immunogenic Factors; Physiological Effects of Drugs; Virus diseases; Orthomyxoviridae Infections; Infection
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections; Influenza, Human; Orthomyxoviridae Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose of quadrivalent VLP vaccine (Experimental): Biological: A single low dose of quadrivalent VLP vaccine
  Interventions: Biological: Low dose of quadrivalent VLP vaccine
- Medium dose of quadrivalent VLP vaccine (Experimental): A single medium dose of quadrivalent VLP vaccine
  Interventions: Biological: Medium dose of quadrivalent VLP vaccine
- High dose of quadrivalent VLP vaccine (Experimental): A single high dose of quadrivalent VLP vaccine
  Interventions: Biological: High dose of quadrivalent VLP vaccine
- Placebo (Placebo Comparator): A single dose of Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low dose of quadrivalent VLP vaccine — A single low dose of quadrivalent VLP vaccine
  Arms: Low dose of quadrivalent VLP vaccine
Biological: Medium dose of quadrivalent VLP vaccine — A single medium dose of quadrivalent VLP vaccine
  Arms: Medium dose of quadrivalent VLP vaccine
Biological: High dose of quadrivalent VLP vaccine — A single high dose of quadrivalent VLP vaccine
  Arms: High dose of quadrivalent VLP vaccine
Biological: Placebo — A single dose of placebo
  Arms: Placebo

SUMMARY:
A phase I/II trial conducted in a single centre, observer-blind, randomized, dose-ranging, placebo-controlled study to evaluate the safety, tolerability, and immunogenicity of a single intramuscular injection of plant-based Seasonal Quadrivalent VLP Influenza Vaccine administered to healthy adults 18-49 years of age.

A total of one hundred and twenty (120) subjects will be randomized in four (4) groups of 30 subjects to receive one injection of either a low, a medium, or a high dose level of VLP of the quadrivalent VLP influenza vaccine or the placebo preparation (100 millimolar (mM) phosphate buffer + 150 mM sodium chloride (NaCl) + 0.01% Tween 80).

DETAILED DESCRIPTION:
The Phase 1 portion of this study will be a dose escalation, cohort staggering (slow enrollment) for the 3 dose levels (low, medium or high dose level) with a placebo-controlled group:

* Cohort 1: A first cohort of thirteen subjects (13) subjects will be randomized, of these ten (10) will be dosed with the lowest dose of the quadrivalent VLP vaccine and three (3) will receive a placebo. The 7-day safety data after the immunization will be collected and reviewed by the Data and Safety Monitoring Board (DSMB) consisting of the Principal Investigator (PI), the Sponsor's Medical Officer and one external medical expert, prior to permitting immunization with the medium dose level.
* Cohort 2: A second cohort of thirteen subjects (13) subjects will be randomized; of these, ten (10) will be dosed with the medium dose of the quadrivalent VLP vaccine and three (3) will receive a placebo. The 7-day safety data after the immunization will be collected and reviewed by the DSMB, prior to permitting immunization with the highest dose.
* Cohort 3: A third cohort of fourteen subjects (14) subjects will be randomized; of these ten (10) dosed with the high dose of the quadrivalent VLP vaccine and four (4) will receive a placebo. The 7-day safety data after the immunization will be collected and reviewed by the DSMB. If the 7-day post-immunization safety data of this cohort is satisfactory according to the DSMB review, the Phase 2 portion of the study will proceed.

The Phase 2 portion of this study will be an observer-blind, randomized, dose-ranging study of the 3 different vaccine doses or a placebo. Therefore, the remaining 20 subjects per vaccine dose will be dosed with the remaining 20 subjects of the placebo group.

Three (3) and 21 days after immunization, key safety (Day 3) and immunogenicity (Day 21) data will be collected and analyzed. All subjects will be followed for safety until Day 201 (6-month follow up), regardless the phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults, 18 to 49 years of age, inclusive.
2. Healthy as judged by the Investigator or designee and determined by medical history, complete general history/symptom-directed physical examination, vital signs, screening laboratories, and medical history conducted no more than 30 days prior to study vaccine administration.
3. BMI of ≥18 and ≤32.
4. Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
5. Accessible by phone on a consistent basis.
6. Give his/her consent to participate in this study (by signing the ICF). In the opinion of the Investigator, competence and willingness to provide written, informed consent for participation after reading the informed consent form. The subject must have adequate opportunity to discuss the study with an Investigator or qualified designee.
7. If female, have a negative serum pregnancy test result prior to immunization.
8. Female of childbearing potential (except subjects in a same sex relationship), must use an effective birth control for the 28 days prior to immunization and must agree to continue employing adequate birth control measures for at least 60 days post-immunization and must have no plan to become pregnant for at least 60 days post-immunization. Highly effective birth control includes hormonal contraceptives (e.g., injectable, topical [patch], estrogenic vaginal ring, etc.), intra-uterine device (IUD), abstinence (confirmed by Investigator), or male condom plus spermicide. Abstinent subjects should be asked what method(s) they would use, should their circumstances change, and subjects without a well-defined plan should be excluded.

Exclusion Criteria:

1. Presence of significant acute or chronic, uncontrolled medical or neuropsychiatric illness. "Uncontrolled" is defined as:

   1. Requiring a new medical or surgical treatment within one month prior to study vaccine administration;
   2. Requiring a change in medication dosage in one month prior to study vaccine administration due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable);
   3. Hospitalization or an event fulfilling the definition of a serious adverse event within one month prior to study vaccine administration.
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse which, in the Investigator's opinion, would render the subject incompetent to provide informed consent or unable to provide valid safety observations and reporting.
3. Any confirmed or suspected immunosuppressive condition or immunodeficiency including history of human immunodeficiency virus (HIV) infection, Hepatitis B or C, or the presence of lymphoproliferative disease.
4. Presence of any febrile illness, oral temperature of >38.0˚C within 24 hours prior to immunization. Such subjects may be re-evaluated for enrolment after resolution of illness.
5. History of autoimmune disease.
6. Administration of any vaccine (including any other influenza vaccine) within 30 days prior to study enrolment or planned administration within the period from the vaccination up to blood sampling at Day 21 or within 30 days prior to blood sampling at Day 201. Immunization on an emergency basis of a tetanus and diphtheria toxoids adsorbed for adult use (Td) will be allowed provided the vaccine is not administered within two weeks prior to study vaccine administration. Receipt of any other emergency immunizations (e.g., rabies) will result in a case-by-case review by the medical monitor of continued participation.
7. Administration of any adjuvanted or investigational influenza vaccine other than a 'simple' seasonal Trivalent influenza vaccine (TIV) or Quadrivalent influenza vaccine (QIV) within 1 year prior to study enrolment or planned administration prior to the end of this trial (Day 201).
8. Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period. Subjects may not participate in any other investigational or marketed drug study while participating in this study.
9. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone per day, or equivalent for more than 7 consecutive days or for 10 or more days in total, within one month of study vaccine administration, any other cytotoxic or immunosuppressant drug, or any globulin preparation within 3 months of vaccination. Low doses of nasal or inhaled glucocorticoids are allowed.
10. Use of high dose inhaled steroids or oral and parenteral high dose steroid medications. Nasal steroids are allowed.
11. Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications, e.g., low-dose aspirin [≤ 325 mg/day (1 regular adult aspirin) or ≤ 81 mg/day (1 baby aspirin)], and without a clinically apparent bleeding tendency are eligible.
12. History of allergy to any of the constituents of the quadrivalent VLP study vaccine, or to the Phosphate-buffered saline (PBS) (used as placebo).
13. History of severe allergic reactions (including anaphylaxis) to any food, medication or bee sting or previous severe asthma.
14. History of tobacco allergy.
15. Continuous use of anti-histamines in the last 4 weeks prior to immunization or use of anti-histamines 48 hours prior to study immunization.
16. Have a rash, dermatological condition, tattoos, or muscle mass at injection site which may interfere with injection site reaction rating.
17. Have received a blood transfusion within 90 days prior to study vaccination.
18. If female, either known pregnancy or urine beta-human chorionic gonadotropin (β-hCG) test results consistent with pregnancy during the screening period and prior to study vaccine administration on Day 0.
19. Female subjects who are lactating.
20. Any vital sign abnormalities: systolic blood pressure, diastolic blood pressure, resting heart rate not well controlled or according to the Investigator's opinion.
21. Cancer or treatment for cancer within 3 years of study vaccine administration. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible. Persons with treated and uncomplicated basal cell carcinoma of the skin are eligible.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10-08; Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of solicited and unsolicited adverse events post-vaccination. | 21 days after injection
Severity of solicited and unsolicited adverse events post-vaccination. | 21 days after injection
Relationship to vaccination of solicited and unsolicited adverse events post-vaccination. | 21 days after injection

SECONDARY OUTCOMES:
Serum HI response induced in subjects against the vaccine strains | 21 days after injection
  Geometric mean titers (GMTs) of hemagglutination inhibition antibodies
capacity of the quadrivalent VLP vaccine to induce specific and functional antibodies against homologous strains | 21 days after injection
  MN assay
Capacity of the quadrivalent VLP vaccine to induce cross-reactive antibodies against heterologous influenza strains | 21 days after injection
  HI and MN assays

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sheldon, MD, Principal Investigator — Miami Research Associate
Locations (1):
- Miami Research Associates, Miami, Florida, United States

REFERENCES:
- [Result] Pillet S, Aubin E, Trepanier S, Bussiere D, Dargis M, Poulin JF, Yassine-Diab B, Ward BJ, Landry N. A plant-derived quadrivalent virus like particle influenza vaccine induces cross-reactive antibody and T cell response in healthy adults. Clin Immunol. 2016 Jul;168:72-87. doi: 10.1016/j.clim.2016.03.008. Epub 2016 Mar 14. PMID 26987887